CLINICAL TRIAL: NCT03354390
Title: A Phase I Study of HERV-E TCR Transduced Autologous T Cells in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: HERV-E TCR Transduced Autologous T Cells in People With Metastatic Clear Cell Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Loyola University Medical Center (LUMC) (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180012; 18-H-0012
Record Dates: First submitted 2017-11-23; First posted 2017-11-28 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Kidney Cancer
Keywords: genetically modified lymphocytes; tumor antigens; T cell receptor immunotherapy; genomic retroviral elements
MeSH Terms: conditions — Kidney Neoplasms | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Level 1 is 1 x 10^6 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight (Experimental): Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 1 x 10^6 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
  Interventions: Biological: cell infusion
- Level 2 is 5 x 10^6 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight (Experimental): Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 5 x 10^6 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
  Interventions: Biological: cell infusion
- Level 3 is 1 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight (Experimental): Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 1 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
  Interventions: Biological: cell infusion
- Level 4 is 5 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight (Experimental): Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 5 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
  Interventions: Biological: cell infusion

INTERVENTIONS:
Biological: cell infusion — This is a phase 1 trial of HERV-E TCR transduced CD8+/CD34+ T cells in HLA-A*11:01 positive patients with metastatic ccRCC. The study is planned based on a Phase 1 3+3 dose escalation design. The maximum tolerated dose (MTD) is defined as the highest dose at which 0 or 1 patient in six has experienced a dose limiting toxicity (DLT). Patients with evaluable advanced/metastatic ccRCC will be recruited in up to 4 dose levels.

SUMMARY:
Background:

Gene transfer is a new cancer therapy takes white blood cells from a person and grows them in a lab. The cells are changed with a virus to attack tumor cells, then returned to the person. Researchers want to see if this therapy fights kidney cancer cells.

Objective:

To see if gene transfer is safe and causes tumors to shrink.

Eligibility:

People at least 18 years old with certain kidney cancer

Design:

Participants will be screened with blood and urine tests. They may have:

* Scans
* Heart, lung, and eye tests
* Lab tests
* Tumor samples taken

Participants will have leukapheresis. Blood will be removed by a needle in an arm. It will go through a machine that removes white blood cells. Plasma and red cells will be returned through a needle in the participant s other arm.

Participants cells will be grown in the lab and genetically changed.

Participants will stay in the hospital 2-3 weeks. There they will:

* Get 2 chemotherapy drugs by catheter (thin plastic tube) inserted into a vein in the chest.
* Get the changed cells via catheter.
* Get a drug to increase white blood cell count and one to make the cells active.
* Recover for about a week.
* Have lab and blood tests.

After leaving the hospital, participants will:

* Take an antibiotic for several months.
* Have leukapheresis.
* Have one- or two-day clinic visits every few weeks for 2 years, and then as determined by their doctor. These will include blood and lab tests, imaging studies, and physical exam.

Participants will have follow-up checks for up to 15 years.

DETAILED DESCRIPTION:
Metastatic renal cell carcinoma (RCC) is an incurable condition. Current therapy for this disease consists of the serial administration of agents such as VEGF, mTOR inhibitors and immunotherapy (high-dose (HD) IL-2 or immune-checkpoint inhibitors). Long-term survival can be achieved with high-doses IL-2 or immune-checkpoint inhibitors. However, of those patients treated with immunotherapy, three quarters will not respond at all and only 5-8% will achieve a complete and durable response.

Allogeneic hematopoietic stem cell transplantation is also capable of inducing prolonged disease regression in patients with metastatic clear cell RCC (ccRCC). In vitro studies have established that transplanted donor T-cells targeting antigens expressed on RCC cells mediate these anti-tumor effects. However, hematopoietic stem cell transplantation can be toxic and associated with a 10-20% risk of procedure-related mortality. The observation that transplanted donor T-cells have the potential to cure a subset of patients with metastatic disease forms the basis for continued efforts in our laboratory to harness the power of T-cells to cure this disorder.

Our team isolated a tumor-specific cytotoxic T lymphocyte (CTL) line from peripheral blood mononuclear cells (PBMCs) obtained after an allogeneic transplant from a patient who showed prolonged tumor regression. Using limiting dilution cloning, we identified an allogeneic (derived from the stem cell donor) CD8+ T-cell clone that killed ccRCC cells in an HLA A11 restricted fashion. Using cDNA expression cloning, we identified a HERV-E derived antigen expressed in the patient s ccRCC cells to be the target of this T-cell clone. Remarkably, we found this HERV-E was expressed in the majority of ccRCC cells with no expression in normal tissues. Based on the identification of the antigenicity of the HERV-E transcripts in ccRCC, our team in collaboration with Dr. Nishimura s laboratory (Loyola University Cardinal Bernardin Cancer Center) has cloned, expressed and characterized the TCR from this CD8+ T-cell clone that recognizes an HLA A11 restricted HERV-E antigen.

This research protocol is therefore designed to evaluate the safety and effectiveness of infusion of HERV-E TCR transduced CD8+/CD34+ enriched T cells in HLA-A*11:01 positive patients with metastatic clear cell RCC. Subjects will receive a novel non-myeloablative immunosuppressive conditioning regimen of cyclophosphamide and fludarabine followed by an infusion of HERV-E TCR transduced CD8+/CD34+ enriched T cells. To mediate T cell survival and sustain function, moderate-doses of IL-2 (aldesleukin) will be administered intravenously twice a day for 14 doses.

The primary endpoint is safety by day 21. Secondary endpoints will include overall response rate, progression-free survival and overall survival. Exploratory studies will include persistence of circulating HERV-E TCR transduced CD8+/CD34+ enriched T cells, changes in immune cell subsets and activation status of T cells, as well as, other immunologic determinants with clinical outcomes at baseline, at different time points during treatment and at the time of disease progression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed RCC with clear-cell component by the Laboratory of Pathology of the NIH and/or outside Pathology Department prior to entering this study.
* Patients must be HLA-A 11:01 positive (confirmed by HLA typing at the NIH DTM)
* Patients must have measurable disease per RECIST version 1.1 and have disease progression during or after the last treatment regimen and within 6 months before study enrollment
* Patients must have received at least one antiangiogenic drug and an immune-checkpoint inhibitor (i.e. nivolumab) unless the patient has contraindications to receiving these medications, the agents are not available to the patient, or the patient declines to receive these drugs due to personal preference.
* Patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 180 days (female patients) or 90 days (male patients) after the end of the treatment if sexually active and able to bear or beget children. In addition, male patients must refrain from sperm donation for 90 days after the final dose of investigational product. Female patients must refrain from egg cell donation for 180 days after the final dose of investigational product
* Patients must be between the ages of 18 and 75 years.
* Patient must have an anticipated life expectancy of at least 3 months.
* Patients must have a performance status of 0 or 1 ECOG performance status (PS) scale.
* Patients must have a caregiver willing to stay with them during the first month of treatment (30 days +/- 7 days).
* Patients receiving treatment with bisphosphonates or denosumab are eligible for enrollment if on a stable dose for greater than or equal to 4 weeks
* Serology:

  * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Organ Function

  * Hematology
  * Absolute neutrophil count greater than or equal to 500/ microL
  * WBC greater than or equal to 1500/microL
  * Platelet count greater than or equal to 75.000/microL (without transfusional support
  * Chemistry
  * Serum AST/ALT less than or equal to 2.5 x upper limit of normal (ULN)
  * Total bilirubin less than or equal to 1.5 mg/dl except for patients with Gilbert s syndrome who must have a total bilirubin less than or equal to 3 mg/dl
  * Creatinine clearance greater than or equal to 50 ml/min/1.73m^2 by the method of CKI-EPI or >=50 ml/min by the method of 24h Clearence of Creatinine Calculation
  * INR < 1.5
  * Cardiology
  * Estimated left ventricular ejection fraction by echocardiography greater than or equal to 45%
  * Respiratory
  * Predicted DLCO / Alveolar Volume Adjusted by PFT >= 45%

EXCLUSION CRITERIA:

* Patients that require immediate therapy due to tumor mass effects or spinal cord compression.
* Patients must not have had standard of care anti-VEGFR therapy (mean half-life around 30 hours), mTOR inhibitors (mean half-life around 30 hours), at least for the last 7 days prior to T-cell infusion and radiotherapy, or major surgery within the last 2 weeks prior to T-cell infusion. For PD-1/PD-L1 inhibitors or CTLA-4 inhibitors, a 4-week period must have elapsed before T-cell infusion. For recent experimental therapies a 28-day period must have elapsed before infusing expanded T-cells.
* Patients with active CNS involvement by malignancy either by imaging or cerebrospinal fluid involvement or biopsy-proven (due to poor prognosis and potential for neurological dysfunction that would confound evaluation of neurological and other adverse events) except for:

  1. Patients with 3 or fewer brain metasteses of <1cm treated with either stereotactic or gamma knife radiotherapy and remained stable on MRI for 2 weeks are eligible.
  2. Patients with surgically resected brain metastases and no evidence of active disease in the CNS at the time of screening evaluation are eligible.
* Patients with hypercalcemia (>10 mg/dL) of malignancy.
* Any prior Grade greater than or equal to 3 immune-related adverse event (irAE) while receiving immunotherapy, including anti-CTLA4 treatment that requires long-term immunosuppressive therapy. Note: Active or history of vitiligo or hypothyroidism will not be a basis for exclusion.
* Patients with second malignancies in addition to their clear cell RCC are not eligible if the second malignancy has required systemic treatment within the past 4 years or is not in complete remission. There are exceptions to this criterion: successfully treated non-metastatic basal cell, squamous cell skin carcinoma, in situ non-invasive cervical cancer and in situ non-invasive breast cancer.
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active coagulation disorders or other major uncontrolled medical illnesses of the respiratory, endocrine, renal, gastrointestinal, genitourinary or immune system, uncontrolled systemic infection, active obstructive or restrictive pulmonary disease.
* Patients who have recent history of cerebrovascular accident, transient ischemic attack should be cleared by the neurology consult service before enrolling this study.
* Patients who have recent history of coronary artery disease or cardiac arrhythmia should be cleared by the cardiology consult service before enrolling this study.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Patients with autoimmune diseases such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis or pancreatitis, and systemic lupus erythematosus that requires treatment with chronic immunosuppressive therapy.
* Systemic corticosteroid steroid therapy of any dose is not allowed within 2 days prior to enrollment.
* The following are exceptions to this criterion:

  * Intranasal, inhaled, and topical steroids
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Unable to understand the investigational nature of the study or give informed consent and does not have a legally authorized representative or surrogate that can provide informed consent.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2026-03-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time of publication or by the end of the protocol, whichever comes first, and available indefinitely.
Access Criteria: Data will be shared through Figshare, which is an open access repository.

REFERENCES:
- [Derived] Barisic S, Brahmbhatt EM, Cherkasova E, Spear TT, Savani U, Pierre S, Scurti GM, Chen L, Igboko M, Nadal R, Zeng G, Parry G, Stroncek DF, Highfill S, Dalheim AV, Reger R, Nishimura MI, Childs RW. Regression of renal cell carcinoma by T cell receptor-engineered T cells targeting a human endogenous retrovirus. J Immunother Cancer. 2024 Sep 11;12(9):e009147. doi: 10.1136/jitc-2024-009147. PMID 39266213
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-H-0012.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight: Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 1 x 10^6 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
- Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight: Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 5 x 10^6 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
- Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight: Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 1 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
- Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight: Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 5 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
Period: Level 1
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Started | 3 | 0 | 0 | 0
Treatment Completed | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Level 2
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Started | 0 | 4 | 0 | 0
Treatment Completed | 0 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 4 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Level 3
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Started | 0 | 0 | 3 | 0
Treatment Completed | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0
Period: Level 4
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Started | 0 | 0 | 0 | 7
Completed Treatment | 0 | 0 | 0 | 7
Completed | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 3
Not completed — Death | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Total
Number analyzed (Participants) | 3 | 4 | 3 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 3 | 6 | 16
  >=65 years | 0 | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2 | 4
  Male | 3 | 3 | 2 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 2 | 3 | 3 | 6 | 14
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 3 | 6 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events at Least Possible Attributed to Treatment Regime for Each Dose Level Using the Common Terminology Criteria for Adverse Events Version 5.0 Except for Hematological Toxicities
Description: Toxicity profile at least possible attributed to treatment regime for each dose level using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 except for hematological toxicities
  Toxicity profile as measured by using the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) for grade 2 and above. According to https://ctep.cancer.gov/, CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. CTCAE grades are defined as:
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
Time Frame: 21 days
Population: Analysis includes all participants that received HERV-E TCR transfused T-cells. Two participants did not receive the HERV-E TCR transfused T-cells because of fast clinical deterioration prior to treatment.
Measure: Number; unit: Adverse events
Groups:
- Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight: Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 5 x10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Number analyzed (Participants) | 3 | 3 | 3 | 6
Adverse events
  Grade 2 (maculopapular rash) | 1 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate Based on the Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline (Version 1.1)
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The participant's best response assignment will depend on the achievement of both measurement and confirmation criteria.
  Partial Response (PR): > 30% decrease in SUL peak; minimum 0.8 unit decrease. Verification with follow-up study if anatomic criteria indicate disease progression.
  Progressive Disease (PD): > 30% increase in SUL peak (minimum 0.8 unit increase in SUL peak), > 75% increase in TLG of the 5 most active lesions, Visible increase in extent of FDG uptake, or new lesions. Verification with follow-up study if anatomic criteria indicate complete or partial response.
  Stable Disease (SD): Does not meet other criteria.
Time Frame: Baseline until date of first documented disease progression or date of death from any cause, whichever comes first, assessed up to Day 127
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants
  Stable Disease | 2 | 0 | 0 | 2
  Progressive Disease | 1 | 3 | 3 | 3
  Partial Response | 0 | 0 | 0 | 1

3. Secondary Outcome: Overall Duration of Response (Days) Based on the Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline (Version 1.1)
Description: Overall duration of response (days) based on the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
  The duration of overall response is measured from the time measurement criteria are met for Complete Response or Partial Response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Baseline until date of first documented response assessed up to Day 127
Population: Analysis includes all participants that received HERV-E TCR transfused T-cells and had either complete response or partial response. Two participants did not receive the HERV-E TCR transfused T-cells because of fast clinical deterioration prior to treatment.
Measure: Number; unit: Days
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Number analyzed (Participants) | 0 | 0 | 0 | 1
Days |  |  |  | 127

4. Secondary Outcome: Median In Weeks to Progression-free Survival
Description: Median in weeks of Progression-free survival. Progression-free survival is defined as from the time of initiation of treatment to the occurrence of disease progression or death, whichever occurs first.
  Disease progression is defined using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (RECIST 1.1), at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Baseline up to Day 192
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight; Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight: Participants with Metastatic Clear Cell Renal Cell Carcinoma will receive a lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by an infusion of 1 x 10^7 HERV-E TCR transduced CD8+/CD34+ enriched T-cells per kg body weight. Following infusion of HERV-E T-cells, participants will receive IL-2 (aldesleukin) which will be administered intravenously twice a day for 14 doses.
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
Number analyzed (Participants) | 3 | 3 | 3 | 6
weeks | 12.9 [8 to 15.5] | 4.4 [4.3 to 8.6] | 4.0 [3.8 to 6.6] | 10.9 [4.6 to 16.2]

5. Secondary Outcome: Median Overall Survival
Description: Median Overall Survival. Overall survival is defined as the
Time Frame: ongoing
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: Up to 5.7 years
Description: Adverse events of any grade will be collected during the first year after cell infusion or until a subject is determined to have disease progression, at which time, the subject will remain on study only for gene therapy related long-term follow up. After one year, or after a subject is determined to have disease progression, no adverse events will be collected, unless they are thought to be at least possibly related to cell infusion.
Arm/Group | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/4 | 1/3 | 3/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 0/3 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4 | 3/3 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=3) | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=4) | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=3) | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=7)
Volume overload (Cardiac disorders) | 1 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Back pain (General disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperkalemia (Investigations) | 0 | 1 | 0 | 0
Hyponatremia (Investigations) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Level 1: 1 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=3) | Level 2: 5 x 10^6 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=4) | Level 3: 1 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=3) | Level 4: 5 x 10^7 HERV-E TCR Transduced CD8+/CD34+ Enriched T-cells Per kg Body Weight (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 2 | 2 | 4
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 3
Alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 3
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1
R submandibular lymph node (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1 | 1
Blood prolactin abnormal (Investigations) | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0 | 0
Bruising (Vascular disorders) | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 2 | 2 | 3 | 2
Abnormal EKG (Cardiac disorders) | 0 | 0 | 0 | 1
BNP increased (Cardiac disorders) | 0 | 0 | 0 | 1
volume overload (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac troponin I increased (Cardiac disorders) | 0 | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 3 | 2 | 3 | 6
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 3 | 3 | 2 | 6
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
CPK increased (Investigations) | 0 | 0 | 1 | 1
Creatinine increased (Investigations) | 1 | 3 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Delirium (Nervous system disorders) | 0 | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Dizziness (General disorders) | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 2 | 1 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 2 | 2 | 1
Febrile neutropenia (General disorders) | 0 | 3 | 2 | 4
Fever (General disorders) | 2 | 2 | 2 | 6
Flushing (General disorders) | 1 | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Generalized edema (General disorders) | 0 | 0 | 1 | 0
GGT increased (Investigations) | 1 | 1 | 0 | 0
Headache (General disorders) | 0 | 1 | 1 | 2
Heart failure (Cardiac disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypercalcemia (Investigations) | 1 | 1 | 2 | 3
Hyperglycemia (Investigations) | 0 | 1 | 0 | 0
Hyperhidrosis (General disorders) | 1 | 1 | 0 | 1
Hyperkalemia (Investigations) | 2 | 0 | 0 | 2
Hypermagnesemia (Investigations) | 1 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hyperphosphatemia (Investigations) | 0 | 2 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hyperuricemia (Investigations) | 1 | 0 | 1 | 2
Hypoalbuminemia (Investigations) | 2 | 2 | 2 | 6
Hypocalcemia (Investigations) | 1 | 1 | 1 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalemia (Investigations) | 0 | 0 | 1 | 2
Hypomagnesemia (Investigations) | 0 | 1 | 1 | 0
Hyponatremia (Investigations) | 3 | 3 | 1 | 6
Hypophosphatemia (Investigations) | 0 | 2 | 2 | 4
Hypotension (Vascular disorders) | 2 | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Blister (Infections and infestations) | 0 | 0 | 0 | 1
INR increased (Investigations) | 1 | 0 | 0 | 0
Insomnia (General disorders) | 1 | 1 | 0 | 1
Blood urea nitrogen increased (Investigations) | 0 | 1 | 0 | 0
Creatine kinase decreased (Investigations) | 1 | 0 | 0 | 0
CRP increased (Investigations) | 0 | 0 | 0 | 2
high ferritin (Investigations) | 0 | 0 | 0 | 1
IgM decreased (Investigations) | 0 | 0 | 1 | 0
Immunoglobulins decreased (IgG and IgA) (Investigations) | 0 | 0 | 0 | 1
Lactate dehydrogenase decreased (Investigations) | 1 | 0 | 0 | 0
Total protein decreased (Investigations) | 1 | 0 | 1 | 2
Total protein increased (Investigations) | 0 | 0 | 0 | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 3 | 3 | 3 | 6
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 3
Neutrophil count decreased (Investigations) | 3 | 3 | 3 | 6
Non-cardiac chest pain (General disorders) | 2 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 3 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 1 | 3 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 3
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2
Syndrome of inappropriate antidiuretic hormone secretion (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 2 | 2 | 1 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
rash (papular) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Superficial thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Testosterone deficiency (Endocrine disorders) | 0 | 0 | 1 | 0
Thyroid stimulating hormone increased (Endocrine disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Weight gain (Investigations) | 1 | 1 | 2 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 2 | 2 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03354390/Prot_SAP_000.pdf